CLINICAL TRIAL: NCT03802760
Title: Cerebral Microembolism in Interventional Cardiology Procedures
Brief Title: Cerebral Microembolism in Cardiology
Acronym: ZEMEK
Status: Completed | Type: Observational
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Principal Investigator, Gabor Erdös, Principal Investigator, Insel Gruppe AG, University Hospital Bern
Other Study IDs: 2018-01066
Record Dates: First submitted 2018-10-22; First posted 2019-01-14 (Actual); Last update posted 2022-11-08 (Actual); Status verified 2022-11

CONDITIONS: Cerebral Embolism
MeSH Terms: conditions — Intracranial Embolism | interventions — Ultrasonography, Doppler, Transcranial

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- TAVI patients: Patients undergoing transfemoral TAVI
  Interventions: Device: Transcranial Doppler (TCD) ultrasound measurement
- MitraClip patients: Patients undergoing MitraClip implantation
  Interventions: Device: Transcranial Doppler (TCD) ultrasound measurement
- TricuspidalClip: Patients undergoing TricuspidalClip implantation
  Interventions: Device: Transcranial Doppler (TCD) ultrasound measurement

INTERVENTIONS:
Device: Transcranial Doppler (TCD) ultrasound measurement — Non-invasive measurement of cerebral embolic load and blood flow using TCD

SUMMARY:
During different interventional cardiology procedures we aim to identify cerebral microemboli load. Further we aim to differentiate the quality and the quantity of cerebral microemboli.We will measure cerebral microemboli in different interventional phases, e.g. during valve deployment, rapid pacing, post-implantation.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Interventional cardiology procedure (TAVI, MitraClip, TricuspidalClip)

Exclusion Criteria:

* Allergy to ultrasound gel or materials contained in the TCD probe
* Missing temporal bone window

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing Interventional cardiology procedure (TAVI, MitraClip, TricuspidalClip)
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2018-10-24 (Actual); Primary Completion 2022-02-24 (Actual); Study Completion 2022-11-06 (Actual)

PRIMARY OUTCOMES:
Quality of cerebral microemboli (solid vs. gaseous) | intraoperative phase, expected to be approx. 4 hours
  The quality of cerebral microemboli is measured by Doppler ultrasonography which automatically detects and analyses the Doppler signal coming from the middle cerebral artery. According to the strength of signal reflection, the signal will be qualified as solid or gaseous.

SECONDARY OUTCOMES:
Quantity of cerebral microemboli load | intraoperative phase, expected to be approx. 4 hours
  The quantity of cerebral microemboli is measured by Doppler ultrasonography which automatically register the counts of solid and gaseous emboli.
Cerebral hemispheric differences (left vs. right) | intraoperative phase, expected to be approx. 4 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology and Pain Medicine, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No